CLINICAL TRIAL: NCT00616330
Title: Vaginal Infection Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lumara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBC-302-602-622467
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-02

CONDITIONS: Vulvovaginitis; Vaginitis
MeSH Terms: conditions — Vulvovaginitis; Vaginitis | interventions — clindamycin phosphate; butoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): clindamycin phosphate/butoconazole nitrate
  Interventions: Drug: clindamycin phosphate/butoconazole nitrate
- 2 (Active Comparator): clindamycin phosphate
  Interventions: Drug: clindamycin phosphate
- 3 (Active Comparator): butoconazole nitrate
  Interventions: Drug: butoconazole nitrate

INTERVENTIONS:
Drug: clindamycin phosphate/butoconazole nitrate — semi solid, single dose
  Arms: 1
Drug: clindamycin phosphate — semi solid, single dose
  Arms: 2
Drug: butoconazole nitrate — semi solid, single dose
  Arms: 3

SUMMARY:
This study will evaluate the efficacy and safety of a vaginal product compared with that of other vaginal products in the treatment of vaginal infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of vaginal infection.
* Patients must be post-menopausal, surgically sterilized or using an acceptable form of birth control.

Exclusion Criteria:

* Patients must not have any other infections
* May not be pregnant or nursing
* May not be receiving any other antimicrobial therapies or any medications that would interfere with the outcome of the study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1443 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical symptom resolution. | baseline, 7 to 10 days and 21 to 30 days

SECONDARY OUTCOMES:
Yeast Culture for Candida | baseline, 7 to 10 days and 21 to 30 days
  Negative Yeast Culture for Candida result=response, Positive Yeast Culture for Candida result=no response
Gram stain Nugent score | baseline, 7 to 10 days and 21 to 30 days
  Gram stain Nugent score of less than 4= resolution, Gram stain Nugent score of greater than 4= no resolution
Saline wet mount for clue cells | baseline, 7 to 10 days and 21 to 30 days
  Saline wet mount negative for clue cells=resolution, Saline wet mount positive for clue cells=no resolution

CONTACTS AND LOCATIONS:
Overall Officials: Jim Joffrion, Study Director — Lumara Health, Inc.
Locations (132):
- United States (81):
  - Clinical Research Consultants, Inc, Birmingham, Alabama
  - Jefferson Clinic, PC, Birmingham, Alabama
  - Choice Research, LLC, Enterprise, Alabama
  - Star W. Research, Chandler, Arizona
  - Precision Trials, LLC/Desert West OB/GYN, Glendale, Arizona
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials LLC, Phoenix, Arizona
  - Visions Clinical Research - Tucson, Tucson, Arizona
  - NEA Women's Clinic, Jonesboro, Arkansas
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - The Woman's Clinic, P.A., Little Rock, Arkansas
  - Precision Clinical Research, Searcy, Arkansas
  - Med Center, Carmichael, California
  - Universal Biopharma Research Institute, Inc./Alta Family Health Clinic, Inc., Dinuba, California
  - Sierra Medical Research, Fresno, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - San Diego Clinical Research Center, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Red Rocks OB/GYN, Lakewood, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Women's Health Care Associates, PC, Hartford, Connecticut
  - Greater Hartford Womens Association/Women's Health, West Hartford, Connecticut
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Insignia Clinical Research, Tampa, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Atlanta Medical Research Institute, Alpharetta, Georgia
  - AMR Research Associates, Bogart, Georgia
  - Medical Network for Educators and Research, Decatur, Georgia
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Atlanta West Women's Center, Douglasville, Georgia
  - The Woman's Clinic, Boise, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Womans Health Practice, LLC, Champaign, Illinois
  - Northern Indiana Womens Health Research, South Bend, Indiana
  - Clinical Trials Management, Mandeville, Louisiana
  - Regional Research Specialists, LLC, Shreveport, Louisiana
  - New England Center for Clinical Research, Inc., Fall River, Massachusetts
  - Activmed Practices & Research, Inc., Haverhill, Massachusetts
  - Healthcare for Women, New Bedford, Massachusetts
  - Female Pelvic Medicine and Urogynecology Institute of Michigan, Grand Rapids, Michigan
  - Women's Health Care Specialists, PC, Paw Paw, Michigan
  - Women's Health Partner, St Louis, Missouri
  - Consultants in Women's Healthcare, St Louis, Missouri
  - New Ballas OB-GYN, Inc., St Louis, Missouri
  - The Medical Group of Northern Nevada, Reno, Nevada
  - Suffolk Ob/Gyn, Port Jefferson, New York
  - Preferred OB/GYN/ Women's Health, Woodbury, New York
  - Eastowne OB-GYN and Infertility, Chapel Hill, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Valaores & Lewis Obstetrics & Gynocology, Winston-Salem, North Carolina
  - Mid Dakota Clinic Center for Women, Bismarck, North Dakota
  - Complete Healthcare for Women, Columbus, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Holzer Clinic, Gallipolis, Ohio
  - Pacific Women's Center, LLC, Eugene, Oregon
  - Medford Women's Clinic, LLP, Medford, Oregon
  - Laurel Highlands Ob/Gyn, PC, Hopwood, Pennsylvania
  - Clinical Trials Research Services, LLC, Natrona Heights, Pennsylvania
  - Associates Ob/Gyn, Germantown, Tennessee
  - Women's Care Center, PLC, Memphis, Tennessee
  - Women Partners in Health, Austin, Texas
  - Advanced Research Associates, Corpus Christi, Texas
  - Research Across America, El Paso, Texas
  - Planned Parenthood of Houston, Houston, Texas
  - The Woman's Hospital of Texas Clinical Research Center, Houston, Texas
  - TMC Life Research, Inc, Houston, Texas
  - Bexar Clinical Trials, LLC, Irving, Texas
  - Willowbend Health and Wellness, Plano, Texas
  - InVisions Consultants, LLC c/o Northeast Ob/Gyn, San Antonio, Texas
  - King's Daughter Clinic, Temple, Texas
  - Tanner Clinic, Layton, Utah
  - Mt. Timpangos Women's Healthcare, Pleasant Grove, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Salt Lake Women's Center, Sandy City, Utah
  - Tidewater Clinical Research, Inc, Virginia Beach, Virginia
  - Walla Walla Clinic, Walla Walla, Washington
  - Hyperion Clinical Research, LLC, Charleston, West Virginia
  - Aurora Advanced Healthcare, Inc, Milwaukee, Wisconsin
- India (21):
  - Institute of Kidney Disease and Research Centre, Ahmedabad, Gujarat
  - Krishna Hospital Surgical & Maternity 201/2/3 Suryadeep Complex, Vadodara, Gujarat
  - Father Muller Medical College Hospital, Mangalore, Kamataka
  - Neha Prakash Hospital, Bangalore, Karnataka
  - KMC Hospital, Mangalore, Karnataka
  - Yenepoya Medical College and Hospital, Mangalore, Karnataka
  - Om Women's Hospital, Nagpur, Maharashtra
  - Avanti Institute of Cardiology, Nagpur, Maharashtra
  - Nagpur Test Tube Baby Centre, Nagpur, Maharashtra
  - VSG Healthcare, Dr. Ganorkar Hospital, Nashik, Maharashtra
  - Nivedita Hospital, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Dr. D. Y. Patil Medical College & Hospital, Pune, Maharashtra
  - Sri Ramachandra Medical College, Chennai, Tamil Nadu
  - Chopra Nursing and Maternity Home, Agra
  - Yashoda Super Speciality Hospital, Ghaziabad
  - Government Maternity Hospital, Hyderabad
  - Makker Medical Center, Lucknow
  - M.K.W. Hospital and Research Centre, New Delhi
  - Sri Ramachandra Medical College, Tamil Nadu
- Ponce School of Medicine, Ponce, Puerto Rico
- Russia (29):
  - Dermatovenerologic Dispensary, Korolyov, Moscow Oblast
  - D.O. Ott Research Institute of Ob/Gyn--Family Planning and Female Health Center, Mendeleevskaya Line, Sankt-Peterburg
  - D.O. Ott Research Institute of Ob/Gyn--Gynecologic Endocrinology, Mendeleyevskaya, Sankt-Peterburg
  - Orkli, LLC, V.o., Sankt-Peterburg
  - Smolensk State Medical Academy of Roszdrav, Smolensk, Smolensk Oblast
  - Kaluga Regional Dermatovenerologic Dispensary, Kaluga
  - Moscow Regional Research Insitute of Obstetrics and Gynecology, Moscow
  - Dermatovenerologic Dispensary #15, Moscow
  - Family Planning and Reproductive Centre, Moscow
  - The Peoples' Friendship University of Russia, Moscow
  - City Clinical Hospital #52, Moscow
  - City Clinical Hospital #31, Moscow
  - Clinic of Skin and Sexual Transmitted Diseases, Moscow
  - City Clinical Hospital #51, Moscow
  - Nizhegorodskiy Dermatovenerologic Scientific Research Institute of Federal Agency for Public Health and Human Services, Nizhny Novgorod
  - Regional Dermatovenerologic Dispensary, Rostov-on-Don
  - Ryazan Regional Clinical Dermatovenerologic Dispensary, Ryazan
  - Juventa--Reproductive Health, Saint Petersburg
  - Medical Mycology Scientific Research Institute at St. Petersburg Medical Academy of Postgraduate Studies of Roszdrav, Saint Petersburg
  - 442 District Military Clinical Hospital of Leningradsky Military District, Saint Petersburg
  - City Dermatovenerologic Dispensary, Saint Petersburg
  - S.M. Kirov Military Medical Academy, MoD of the Russian Federation, Saint Petersburg
  - L.G. Sokolov Clinical Hospital #122 of the Federal Medical-Biologic Agency--#321, Saint Petersburg
  - L.G. Sokolov Clinical Hospital #122 of the Federal Medical-Biologic Agency--#322, Saint Petersburg
  - Leningradskiy Regional Clinical Hospital, Saint Petersburg
  - Family Planning and Reproductive Centre, Saint Petersburg
  - St. Petersburg State I.I. Mechnikov Medical Academy of Roszdrav, Saint Petersburg
  - Andros Clinic, LLC, Saint Petersburg
  - Smolensk Dermatovenerologic Dispensary, Smolensk